CLINICAL TRIAL: NCT03582358
Title: Evaluation of a Strategy for the Presentation of Oral Nutritional Supplements (ONS) in Verrines for Managing Undernutrition in the Elderly Undergoing Follow-up Care and Geriatric Rehabilitation. Biomedical, Monocentric, Comparative, Clustered and Open Randomized Research Study
Brief Title: Evaluation of a Strategy for the Presentation of Oral Nutritional Supplements in Verrines for Managing Undernutrition in the Elderly Undergoing Follow-up Care and Geriatric Rehabilitation
Acronym: VERRINES-CNO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VAN WYMELBEKE Lactalis 2017
Record Dates: First submitted 2018-06-07; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Patients Hospitalized in Follow up Care or Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Verrine: Patients served verrines
  Interventions: Other: Food weighing
- CNO: Patients served wrapped supplements
  Interventions: Other: Food weighing

INTERVENTIONS:
Other: Food weighing — Quantification of food intake over three consecutive days (D5, D6 and D7 then D26, D27 and D28) by weighing the food served and the leftovers at and after mealtimes.

SUMMARY:
Protein-energy malnutrition results from an imbalance between the body's intake and needs. Among the elderly in long-term care, the prevalence of undernutrition varies from 30% to 70%. It is responsible for or aggravates a state of fragility or dependence, and promotes the occurrence of morbidities. It is also associated with worsening prognosis for underlying diseases and increases the risk of death. Nutritional management of undernutrition is an issue, especially in health facilities. Among the various existing nutritional care methods, oral nutritional supplements should be considered in the event of failure of food enrichment measures or even at the outset in undernourished elderly people. However, compliance or acceptance of these products among the elderly remains limited and variable with consumption of oral nutritional supplements ranging between 48% and 94% according to studies, and, because of their ease of prescription, oral supplements are sometimes the only nutritional intervention.

ELIGIBILITY:
Inclusion Criteria:

* Undernourished or at-risk individuals with blood albumin levels below 35 g/L or prealbumin levels below 200 mg/L,
* Person admitted to geriatric follow up care less than 48 hours ago,
* Person fed orally,
* Person with a prescription for an ONS,
* Person who speaks and understands French.

Exclusion Criteria:

* Person not affiliated to a national health insurance scheme
* Person requiring enteral or parenteral feeding
* Person refusing to consume ONS
* People at the very end of their lives

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Quantity of oral nutritional supplements consumed daily | through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France